CLINICAL TRIAL: NCT01091025
Title: A Comparative Analysis of the Clinical Efficacy of Two Approaches in the Screening for Cystic Fibrosis Related Diabetes in Adult With Cystic Fibrosis: i) a Selective Approach; ii) an Unselected Annual Oral Glucose Tolerance Test
Brief Title: Comparing Two Different Approaches in the Screening of Cystic Fibrosis Related Diabetes
Acronym: CFRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CRO-1210
Record Dates: First submitted 2010-03-18; First posted 2010-03-23 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2010-03

CONDITIONS: Screening of Cystic Fibrosis Related Diabetes
Keywords: Adults; Cystic Fibrosis Related Diabetes; Screening; Oral glucose tolerance test; Royal Brompton & Harefield Foundation Trust

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CF patients without known diagnose of CFRD (Other): There is only one arm. All patients in the study had the same procedures (ie. an OGTT). Investigators used the screening criteria in parallel to this.
  Interventions: Other: Glucose profile for 2 weeks

INTERVENTIONS:
Other: Glucose profile for 2 weeks — A study subject has an abnormal OGTT will be referred to a cystic fibrosis consultant who is not involved in the study.

SUMMARY:
The incidence of cystic fibrosis related diabetes (CFRD) has risen significantly as patients' survival improves. Early diagnosis of CFRD is crucial to prevent the unnecessary deterioration of lung function and nutritional status, both of which affect the patient's overall survival. The oral glucose tolerance test (OGGT) is the accepted method for detecting CFRD. The Cystic Fibrosis Trust guidelines (2004) recommend that patients with CF over the age of twelve years should be screened annually. Most hospitals use an annual OGTT. Performing OGTT on all CF patients is inconvenient and may not be cost effective, as patients have to starve overnight and need to spend an extra 2 hours in the hospital in addition to all the other annual review tests. In our centre, a selective approach is used. If patients have an abnormal random blood glucose and /or abnormal glycosylated haemoglobin (HbA1c) and/or symptoms of hyperglycaemia or unexplained weight loss then an OGTT will be performed.

The aims of this study are

1. To compare the clinical efficiency in the screening for CFRD in the two different methods: i)a selective approach , ii)an unselected annual OGTT for all patients.
2. To compare the cost effectiveness of the two approaches in the screening for CFRD.

DETAILED DESCRIPTION:
CFRD affects 30% of all patients with cystic fibrosis (CF) by the age of twenty-five. Early diagnosis of CFRD is crucial to prevent the unnecessary deterioration of pulmonary function and nutritional status, both of which affect the patient's overall survival. The selective approach takes less patient time and is less expensive. If it is equally accurate it should be used routinely. The oral glucose tolerance test (OGTT) is the accepted method for detecting CFRD and the Cystic Fibrosis Trust guidelines recommend that patients with CF over the age of twelve years should be screened annually. Yung et al, questioned this approach and argued that performing OGTT on all CF patients is inconvenient and may not be cost effective, as patients have to starve overnight and need to spend an extra 2 hours in the hospital in addition to all the other annual review tests.

In this study, a selective approach in performing OGTTs in the screening for CFRD will be used; this includes the use of a combination of clinical and biochemical criteria that of abnormal random blood glucose and /or abnormal glycosylated haemoglobin (HbA1c) and/or symptoms of hyperglycaemia, or weight loss.

ELIGIBILITY:
Inclusion Criteria:

* first one hundred consecutive clinically stable patients with CF attending annual review from January 2009
* 16 years of age and over will be eligible for the study.

Exclusion Criteria:

* patients with an existing diagnosis of CFRD.
* patients with an infective exacerbation (i.e. on a new course of antibiotics)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To identify if using the selective approach to screen for CFRD is as accurate as screening all patients with OGTT at annual review. | 6 months
  1. Patients identified for OGTT based on the selective approach by the two independent reviewers will be compared.
  2. Patients will form two groups:
     i)those identified as needing OGTT, ii)those on whom they considered it unnecessary
  3. The results of the two groups will then be compared with the data obtain from OGTT to which the two reviewers were 'blinded'

SECONDARY OUTCOMES:
Which is the more cost effective way of screening all patients with OGTT? | 6 months
  1. Calculate the cost of glucose powder and laboratory analysis for each OGTT.
  2. Compare the cost effectiveness of carrying out OGTT on patients identified by the selective approach with the cost of carrying out OGTT on all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Maragret E Hodson, Professor, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton & Harefield NHS Foundation Trust, London, United Kingdom